CLINICAL TRIAL: NCT03906617
Title: Title of Project: Liposomal Bupivacaine (Exparel) Versus Bupivacaine And Dexamethasone Intercostal Nerve Blocks For Robotic Thoracic Surgery: A Prospective Randomized Single-Blinded Clinical Trial
Brief Title: Bupivacaine/Epinephrine +Dexamethasone vs. Liposomal Bupivacaine
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Principal Investigator, Kingsuk Ganguly, M.D., Assistant Professor of Anesthesiology, The Cooper Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18039
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Robotic Lung Surgery
MeSH Terms: interventions — Bupivacaine; Epinephrine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bupivacaine/epinephrine + dexamethasone (Experimental)
  Interventions: Drug: Intercostal nerve block and wound infiltration with bupivacaine/epinephrine + dexamethasone
- Liposomal bupivacaine (Active Comparator)
  Interventions: Drug: Intercostal nerve block and wound infiltration with liposomal bupivacaine

INTERVENTIONS:
Drug: Intercostal nerve block and wound infiltration with liposomal bupivacaine — Intercostal nerve block and wound infiltration with liposomal bupivacaine during robotic lung resection surgery. 266mg of liposomal bupivacaine with 24 ml of 0.5% bupivacaine will be used.
  Arms: Liposomal bupivacaine
Drug: Intercostal nerve block and wound infiltration with bupivacaine/epinephrine + dexamethasone — Intercostal nerve block and wound infiltration with liposomal bupivacaine during robotic lung resection surgery. 42 ml of 0.5% Bupivacaine/epinephrine with 8mg dexamethasone will be used.
  Arms: Bupivacaine/epinephrine + dexamethasone

SUMMARY:
This study will assess analgesia after robotic lung surgery. Subjects will be randomized to receive wound infiltration and intercostal nerve block with either liposomal bupivacaine or bupivacaine/epinephrine + dexamethasone. Liposomal bupivacaine is a newer local anesthetic product and has not been compared to a combination of bupivacaine/epinephrine + dexamethasone in the context of pain control after robotic lung surgery.

ELIGIBILITY:
Inclusion Criteria:

* undergoing robotic wedge resection or lobectomy for lung mass(es)

Exclusion Criteria:

* emergency case
* history of opiate abuse
* chronic pain syndrome
* intravenous drug use
* chronic use of oral steroids
* pregnancy
* imprisonment
* body weight lower than 70 kg
* liver failure
* uninsured patients
* non-verbal patients or patients who are unable to rate their pain on a visual analogue pain scale
* history of allergic reaction to any of the drugs used in the study: bupivacaine, liposomal bupivacaine, dexamethasone

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-04-10 (Estimated); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale pain scores | 24 hours post-surgery
  Visual Analogue Scale (VAS) pain score will be assessed for non-inferiority of bupivacaine/epinephrine +dexamethasone vs. liposomal bupivacaine. A non-inferiority margin of 2 points on the VAS scale will be considered non-inferior.

CONTACTS AND LOCATIONS:
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States